CLINICAL TRIAL: NCT05238909
Title: Developing Novel Biomarkers of Plexiform Neurofibroma Tumor Burden
Brief Title: Developing Biomarkers of Plexiform Tumor Burden in Patients With Neurofibromatosis-Type 1
Status: Enrolling by invitation | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Carlos Prada, MD, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2022-4928; 7R61NS122094-02 (NIH); 4R33NS122094-03 (NIH)
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Neurofibromatosis 1; NF1; Neurofibromatosis Type 1
Keywords: NF1; Plexiform neurofibromas; neurofibromatosis type 1; neurofibromas
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Neurofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood plasma, DNA, and RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify tumor biomarkers in individuals with Neurofibromatosis type 1 (NF1). Biomarkers are signals that the investigator can measure that tell us about a process such as progress of a disease or treatment. Individuals with this diagnosis are at an elevated risk of developing a type of tumor called a plexiform neurofibroma. Currently, detecting the risk factors of these tumors in children is difficult and requires whole body imaging. The NF1 team at Lurie Children's established a way of using blood plasma in mice with neurofibromatosis type 1 to identify biomarkers that might signal the presence of tumors in people with NF1.

This study is an effort to create biomarker profiles of patients with NF1 with known tumors. The study team will utilize whole-body MRI and mass spectrometry (a method for identifying unknown compounds and the properties of molecules). The ultimate goal of this study is to better understand the tumor biomarkers in patients with NF1.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a common inherited human disorder, with a frequency of approximately 1:2500 worldwide. A hallmark of NF1 is development of plexiform neurofibromas (PNFs) in 30 to 50% of NF1 patients. Currently, there are no biomarkers of tumor burden and whole-body magnetic resonance imaging (MRI) is expensive and limited to few centers. The investigator established an unbiased pipeline to identify candidate biomarker signals of tumor burden using plasma from neurofibroma-bearing DhhCre;Nf1fl/fl mice using untargeted metabolomics. Our preliminary data show that glucosylceramide (GC) is the most significantly deregulated compound in plasma from neurofibroma-bearing DhhCre;Nf1fl/fl mice. The investigator developed a novel targeted mass spectrometry method to accurately quantify multiple elevated GC and lactosylceramide (LC) species. In this proposal, the investigator will combine the clinical infrastructure of the NF1 comprehensive program and advance imaging at Ann & Robert H. Lurie Children's Hospital of Chicago with the mass spectrometry capabilities at Cincinnati Children's Hospital Medical Center.

Taking advantage of our large, well-characterized, Lurie Children's NF1 population, the investigator propose to perform analytical validation studies of candidate GC/LC biomarker signature of tumor burden in plasma from NF1 patients with defined numbers of PNF (tumor burden) by whole body MRI. The potential outcomes of our study are identification of candidate biomarker of tumor burden that contribute to patient risk stratification, and analytical validation of GC/LC biomarker signature (context of use). Collectively, this work represents a synergistic approach for discovery and validation of biomarkers of tumor burden in NF1.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with known diagnosis of neurofibromatosis type 1 (NF1)

Exclusion Criteria:

1. Patient does not meet NF1 diagnostic criteria
2. Mosaic NF1 individuals
3. Pregnant at Screening
4. Patients who do not have the ability/capacity to undergo the informed consent process OR whose parent/legal guardian is unable to undergo the informed consent process.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the NF1 Clinical Program at Lurie Children's Hospital of Chicago
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Determine if glucosylceramide (GC) and lactosylceramide (LC) species levels correlate with tumor burden in patients with NF1 | 1 year
  The investigator and team will collect blood samples from individuals with NF1 stratified plexiform tumor (PNF) burden (none, small, intermediate, and large) versus age and sex matched healthy control.
Test if tumor burden correlates with GC and LC signature in individuals with NF1 who are undergoing clinical treatment with MEK inhibitors | 1 year
  The investigator and team will enroll 20 individuals with NF1 and inoperable PNFs in treatment with MEK inhibitors to correlate biomarker with tumor burden changes with therapy.
Assemble a longitudinal cohort of individuals with NF1 with plexiform neurofibromas (n=100) for deep phenotyping and tumor burden response to MEK inhibitors | 1 year
  Whole-body MRI at baseline and at time of annual visit (9-to-18-month intervals) will be used to deeply phenotype individuals based on tumor burden and tumor volume. Individuals will undergo plasma collection and clinical history assessment (medications, diet log, supplements, and anthropometric measurements) at each visit. For patients undergoing treatment with MEK inhibitors, a sample prior to treatment will be collected during this study.
Determine if glucosylceramide (GC) and lactosylceramide (LC) signature correlates with plexiform neurofibroma burden change in longitudinal cohort of 100 individuals with PNFs | 1 year
  The investigator and team will test GC/LC levels using validated mass spectrometry target method for quantification of these biomarkers.
Tumor volumetric analysis will be performed to correlate with GC/LC monitoring biomarker signature | 1 year
  GC/LC biomarker thresholds (cut-off) will be refined to evaluate predictive ability to identify individuals with large tumor burden. Tumor burden will be measured from whole-body MRI analysis with post-imaging processing software.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Prada, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Le LQ, Parada LF. Tumor microenvironment and neurofibromatosis type I: connecting the GAPs. Oncogene. 2007 Jul 12;26(32):4609-16. doi: 10.1038/sj.onc.1210261. Epub 2007 Feb 12. PMID 17297459
- [Background] McCormick F. Ras signaling and NF1. Curr Opin Genet Dev. 1995 Feb;5(1):51-5. doi: 10.1016/s0959-437x(95)90053-5. PMID 7749326
- [Background] Birnbaum RA, O'Marcaigh A, Wardak Z, Zhang YY, Dranoff G, Jacks T, Clapp DW, Shannon KM. Nf1 and Gmcsf interact in myeloid leukemogenesis. Mol Cell. 2000 Jan;5(1):189-95. doi: 10.1016/s1097-2765(00)80415-3. PMID 10678181
- [Background] Bollag G, Clapp DW, Shih S, Adler F, Zhang YY, Thompson P, Lange BJ, Freedman MH, McCormick F, Jacks T, Shannon K. Loss of NF1 results in activation of the Ras signaling pathway and leads to aberrant growth in haematopoietic cells. Nat Genet. 1996 Feb;12(2):144-8. doi: 10.1038/ng0296-144. PMID 8563751
- [Background] Largaespada DA, Brannan CI, Jenkins NA, Copeland NG. Nf1 deficiency causes Ras-mediated granulocyte/macrophage colony stimulating factor hypersensitivity and chronic myeloid leukaemia. Nat Genet. 1996 Feb;12(2):137-43. doi: 10.1038/ng0296-137. PMID 8563750
- [Background] Ratner N, Miller SJ. A RASopathy gene commonly mutated in cancer: the neurofibromatosis type 1 tumour suppressor. Nat Rev Cancer. 2015 May;15(5):290-301. doi: 10.1038/nrc3911. Epub 2015 Apr 16. PMID 25877329
- [Background] Prada CE, Rangwala FA, Martin LJ, Lovell AM, Saal HM, Schorry EK, Hopkin RJ. Pediatric plexiform neurofibromas: impact on morbidity and mortality in neurofibromatosis type 1. J Pediatr. 2012 Mar;160(3):461-7. doi: 10.1016/j.jpeds.2011.08.051. Epub 2011 Oct 11. PMID 21996156
- [Background] Wu J, Williams JP, Rizvi TA, Kordich JJ, Witte D, Meijer D, Stemmer-Rachamimov AO, Cancelas JA, Ratner N. Plexiform and dermal neurofibromas and pigmentation are caused by Nf1 loss in desert hedgehog-expressing cells. Cancer Cell. 2008 Feb;13(2):105-16. doi: 10.1016/j.ccr.2007.12.027. PMID 18242511
- [Background] Jessen WJ, Miller SJ, Jousma E, Wu J, Rizvi TA, Brundage ME, Eaves D, Widemann B, Kim MO, Dombi E, Sabo J, Hardiman Dudley A, Niwa-Kawakita M, Page GP, Giovannini M, Aronow BJ, Cripe TP, Ratner N. MEK inhibition exhibits efficacy in human and mouse neurofibromatosis tumors. J Clin Invest. 2013 Jan;123(1):340-7. doi: 10.1172/JCI60578. Epub 2012 Dec 10. PMID 23221341
- [Background] Jousma E, Rizvi TA, Wu J, Janhofer D, Dombi E, Dunn RS, Kim MO, Masters AR, Jones DR, Cripe TP, Ratner N. Preclinical assessments of the MEK inhibitor PD-0325901 in a mouse model of Neurofibromatosis type 1. Pediatr Blood Cancer. 2015 Oct;62(10):1709-16. doi: 10.1002/pbc.25546. Epub 2015 Apr 22. PMID 25907661
- [Background] Dombi E, Baldwin A, Marcus LJ, Fisher MJ, Weiss B, Kim A, Whitcomb P, Martin S, Aschbacher-Smith LE, Rizvi TA, Wu J, Ershler R, Wolters P, Therrien J, Glod J, Belasco JB, Schorry E, Brofferio A, Starosta AJ, Gillespie A, Doyle AL, Ratner N, Widemann BC. Activity of Selumetinib in Neurofibromatosis Type 1-Related Plexiform Neurofibromas. N Engl J Med. 2016 Dec 29;375(26):2550-2560. doi: 10.1056/NEJMoa1605943. PMID 28029918
- [Background] Dombi E, Solomon J, Gillespie AJ, Fox E, Balis FM, Patronas N, Korf BR, Babovic-Vuksanovic D, Packer RJ, Belasco J, Goldman S, Jakacki R, Kieran M, Steinberg SM, Widemann BC. NF1 plexiform neurofibroma growth rate by volumetric MRI: relationship to age and body weight. Neurology. 2007 Feb 27;68(9):643-7. doi: 10.1212/01.wnl.0000250332.89420.e6. Epub 2007 Jan 10. PMID 17215493
- [Background] Gross AM, Wolters PL, Dombi E, Baldwin A, Whitcomb P, Fisher MJ, Weiss B, Kim A, Bornhorst M, Shah AC, Martin S, Roderick MC, Pichard DC, Carbonell A, Paul SM, Therrien J, Kapustina O, Heisey K, Clapp DW, Zhang C, Peer CJ, Figg WD, Smith M, Glod J, Blakeley JO, Steinberg SM, Venzon DJ, Doyle LA, Widemann BC. Selumetinib in Children with Inoperable Plexiform Neurofibromas. N Engl J Med. 2020 Apr 9;382(15):1430-1442. doi: 10.1056/NEJMoa1912735. Epub 2020 Mar 18. PMID 32187457
- [Background] Fletcher JS, Pundavela J, Ratner N. After Nf1 loss in Schwann cells, inflammation drives neurofibroma formation. Neurooncol Adv. 2019 Nov 22;2(Suppl 1):i23-i32. doi: 10.1093/noajnl/vdz045. eCollection 2020 Jul. PMID 32642730
- [Background] Fletcher JS, Springer MG, Choi K, Jousma E, Rizvi TA, Dombi E, Kim MO, Wu J, Ratner N. STAT3 inhibition reduces macrophage number and tumor growth in neurofibroma. Oncogene. 2019 Apr;38(15):2876-2884. doi: 10.1038/s41388-018-0600-x. Epub 2018 Dec 12. PMID 30542122
- [Background] Prada CE, Jousma E, Rizvi TA, Wu J, Dunn RS, Mayes DA, Cancelas JA, Dombi E, Kim MO, West BL, Bollag G, Ratner N. Neurofibroma-associated macrophages play roles in tumor growth and response to pharmacological inhibition. Acta Neuropathol. 2013 Jan;125(1):159-68. doi: 10.1007/s00401-012-1056-7. Epub 2012 Oct 26. PMID 23099891
- [Background] Fletcher JS, Wu J, Jessen WJ, Pundavela J, Miller JA, Dombi E, Kim MO, Rizvi TA, Chetal K, Salomonis N, Ratner N. Cxcr3-expressing leukocytes are necessary for neurofibroma formation in mice. JCI Insight. 2019 Feb 7;4(3):e98601. doi: 10.1172/jci.insight.98601. PMID 30728335
- [Background] Wu J, Dombi E, Jousma E, Scott Dunn R, Lindquist D, Schnell BM, Kim MO, Kim A, Widemann BC, Cripe TP, Ratner N. Preclincial testing of sorafenib and RAD001 in the Nf(flox/flox) ;DhhCre mouse model of plexiform neurofibroma using magnetic resonance imaging. Pediatr Blood Cancer. 2012 Feb;58(2):173-80. doi: 10.1002/pbc.23015. Epub 2011 Feb 11. PMID 21319287
- [Background] Bujak R, Struck-Lewicka W, Markuszewski MJ, Kaliszan R. Metabolomics for laboratory diagnostics. J Pharm Biomed Anal. 2015 Sep 10;113:108-20. doi: 10.1016/j.jpba.2014.12.017. Epub 2014 Dec 25. PMID 25577715
- [Background] Grissa D, Petera M, Brandolini M, Napoli A, Comte B, Pujos-Guillot E. Feature Selection Methods for Early Predictive Biomarker Discovery Using Untargeted Metabolomic Data. Front Mol Biosci. 2016 Jul 8;3:30. doi: 10.3389/fmolb.2016.00030. eCollection 2016. PMID 27458587
- [Background] Watanabe M, Roth TL, Bauer SJ, Lane A, Romick-Rosendale LE. Feasibility Study of NMR Based Serum Metabolomic Profiling to Animal Health Monitoring: A Case Study on Iron Storage Disease in Captive Sumatran Rhinoceros (Dicerorhinus sumatrensis). PLoS One. 2016 May 27;11(5):e0156318. doi: 10.1371/journal.pone.0156318. eCollection 2016. PMID 27232336
- [Background] Setchell KD, Nardi E, Battezzati PM, Asciutti S, Castellani D, Perriello G, Clerici C. Novel soy germ pasta enriched in isoflavones ameliorates gastroparesis in type 2 diabetes: a pilot study. Diabetes Care. 2013 Nov;36(11):3495-7. doi: 10.2337/dc12-1615. Epub 2013 Jul 8. PMID 23835688
- [Background] Weiss B, Plotkin S, Widemann B, Tonsgard J, Blakeley J, Allen J, Schorry E, Korf B, Rosser T, Goldman S, Vinks A, Cutter G, Dombi E, Ratner N, Packer R, Fisher M. NFM-06. NF106: PHASE 2 TRIAL OF THE MEK INHIBITOR PD-0325901 IN ADOLESCENTS AND ADULTS WITH NF1-RELATED PLEXIFORM NEUROFIBROMAS: AN NF CLINICAL TRIALS CONSORTIUM STUDY. Neuro Oncol. 2018 Jun;20(Suppl 2):i143. doi: 10.1093/neuonc/noy059.514. Epub 2018 Jun 22. PMCID: PMC6012484.
- [Background] Johnson CH, Ivanisevic J, Benton HP, Siuzdak G. Bioinformatics: the next frontier of metabolomics. Anal Chem. 2015 Jan 6;87(1):147-56. doi: 10.1021/ac5040693. Epub 2014 Nov 20. No abstract available. PMID 25389922
- [Background] Redrup MJ, Igarashi H, Schaefgen J, Lin J, Geisler L, Ben M'Barek M, Ramachandran S, Cardoso T, Hillewaert V. Sample Management: Recommendation for Best Practices and Harmonization from the Global Bioanalysis Consortium Harmonization Team. AAPS J. 2016 Mar;18(2):290-3. doi: 10.1208/s12248-016-9869-2. Epub 2016 Jan 28. PMID 26821803
- [Background] van de Merbel N, Savoie N, Yadav M, Ohtsu Y, White J, Riccio MF, Dong K, de Vries R, Diancin J. Stability: recommendation for best practices and harmonization from the Global Bioanalysis Consortium Harmonization Team. AAPS J. 2014 May;16(3):392-9. doi: 10.1208/s12248-014-9573-z. Epub 2014 Feb 19. PMID 24550081
- [Background] Sankoh AJ, Huque MF, Dubey SD. Some comments on frequently used multiple endpoint adjustment methods in clinical trials. Stat Med. 1997 Nov 30;16(22):2529-42. doi: 10.1002/(sici)1097-0258(19971130)16:223.0.co;2-j. PMID 9403954